CLINICAL TRIAL: NCT00930514
Title: A Two Stage Phase Ib Study to Investigate the Pharmacokinetics, Safety and Tolerability of Rituximab Subcutaneous (SC) Formulation in Patients With Follicular Lymphoma (FL) as Part of Maintenance Treatment
Brief Title: A Pharmacokinetic Study of Subcutaneous and Intravenous Rituximab in Participants With Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22333; 2008-008490-60
Record Dates: First submitted 2009-06-16; First posted 2009-06-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

ARMS (6):
- Rituximab IV 375 mg/m^2 (Stage 1: Cohort A) (Active Comparator)
  Interventions: Drug: Rituximab
- Rituximab IV 375 mg/m^2 (Stage 2: Cohort E) (Active Comparator)
  Interventions: Drug: Rituximab
- Rituximab SC 1400 mg (Stage 2: Cohort F) (Experimental)
  Interventions: Drug: Rituximab
- Rituximab SC 375 mg/m^2 (Stage 1: Cohort B) (Experimental)
  Interventions: Drug: Rituximab
- Rituximab SC 625 mg/m^2 (Stage 1: Cohort C) (Experimental)
  Interventions: Drug: Rituximab
- Rituximab SC 800 mg/m^2 (Stage 1: Cohort D) (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab subcutaneous injection at 1400 mg dose level, administered every 2 or 3 months.
  Arms: Rituximab SC 1400 mg (Stage 2: Cohort F)
Drug: Rituximab — Rituximab subcutaneous injection at 800 mg/m^2 dose level, administered every 2 or 3 months.
  Other Names: MabThera/Rituxan
  Arms: Rituximab SC 1400 mg (Stage 2: Cohort F); Rituximab SC 800 mg/m^2 (Stage 1: Cohort D)
Drug: Rituximab — Rituximab subcutaneous injection 625 mg/m^2 administered every 2 or 3 months.
  Other Names: MabThera/Rituxan
  Arms: Rituximab SC 625 mg/m^2 (Stage 1: Cohort C)
Drug: Rituximab — Rituximab intravenous infusion 375 milligram per square meter (mg/m^2) administered every 2 or 3 months.
  Other Names: MabThera/Rituxan
  Arms: Rituximab IV 375 mg/m^2 (Stage 1: Cohort A); Rituximab IV 375 mg/m^2 (Stage 2: Cohort E)
Drug: Rituximab — Rituximab subcutaneous injection 375 mg/m^2 administered every 2 or 3 months.
  Other Names: MabThera/Rituxan
  Arms: Rituximab SC 375 mg/m^2 (Stage 1: Cohort B)

SUMMARY:
This 2 stage study will compare the pharmacokinetics and safety profile of subcutaneous and intravenous rituximab in participants with follicular lymphoma. In the first stage, participants who have achieved at least a partial response after induction treatment with intravenous rituximab will be randomized to one of 3 treatment cohorts, to receive rituximab 375 milligram per square meter (mg/m^2) intravenously, 375 mg/m^2 subcutaneously or 625 mg/m^2 subcutaneously, and pharmacokinetics evaluated on an ongoing basis. Upon selection of the subcutaneous dose (800 mg/m^2) which results in rituximab trough plasma concentration (C trough) values comparable to those achieved with the intravenous formulation, participants in the second stage of the study will be randomized to receive either the subcutaneous or intravenous formulation to demonstrate comparability of the C trough levels with both routes of administration. Maintenance therapy will continue every 2 or 3 months with the subcutaneous formulation.

ELIGIBILITY:
Inclusion Criteria:

* CD20-positive follicular non-Hodgkin's lymphoma (NHL)
* Documented partial or complete response a the end of induction treatment with rituximab
* Must have completed induction treatment, and received at least 1 dose of intravenous rituximab maintenance treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of less than and equal to (<=) 2
* Life expectancy of greater than and equal to (>=) 6 months

Exclusion Criteria:

* Histological evidence of transformation of NHL, or types of NHL other than follicular lymphoma
* Presence or history of central nervous system disease
* History of malignancy other than follicular NHL
* Recent major surgery (within 4 weeks prior to screening), excluding lymph node biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Minimum Observed Plasma Trough Concentration (C trough) | Up to 29 months

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to end of Dosing Interval (AUCtau) | Up to 29 months
Maximum Observed Plasma Concentration (Cmax) | Up to 29 months
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to 29 months
Plasma Decay Half-Life (t1/2) | Up to 29 months
Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Up to 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Rosario
- Australia (4):
  - Kogarah, New South Wales
  - Sydney, New South Wales
  - Kurralta Park, South Australia
  - Fitzroy, Victoria
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - Barretos, São Paulo
  - São Paulo, São Paulo
- Canada (5):
  - Calgary, Alberta
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Montreal, Quebec
  - Québec, Quebec
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Herlev, Denmark
- Ecuador (2):
  - Guayaquil
  - Quito
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- France (3):
  - Marseille
  - Montpellier
  - Reims
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (4):
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
  - Pisa, Tuscany
- Mexico (3):
  - Aguascalientes
  - Mexico City, Distrito Federal
  - Monterrey
- Oslo, Norway
- Lima, Peru
- Poland (2):
  - Warsaw
  - Wroclaw
- Moscow, Russia
- Bratislava, Slovakia
- Seoul, South Korea
- Spain (3):
  - Barcelona, Barcelona
  - Salamanca, Salamanca
  - Seville, Sevilla
- Sweden (4):
  - Huddinge
  - Sundsvall
  - Umeå
  - Uppsala
- Basel, Switzerland
- United Kingdom (4):
  - Cambridge
  - London
  - Manchester
  - Nottingham

REFERENCES:
- [Derived] Salar A, Avivi I, Bittner B, Bouabdallah R, Brewster M, Catalani O, Follows G, Haynes A, Hourcade-Potelleret F, Janikova A, Larouche JF, McIntyre C, Pedersen M, Pereira J, Sayyed P, Shpilberg O, Tumyan G. Comparison of subcutaneous versus intravenous administration of rituximab as maintenance treatment for follicular lymphoma: results from a two-stage, phase IB study. J Clin Oncol. 2014 Jun 10;32(17):1782-91. doi: 10.1200/JCO.2013.52.2631. Epub 2014 May 12. PMID 24821885
- [Derived] Mao CP, Brovarney MR, Dabbagh K, Birnbock HF, Richter WF, Del Nagro CJ. Subcutaneous versus intravenous administration of rituximab: pharmacokinetics, CD20 target coverage and B-cell depletion in cynomolgus monkeys. PLoS One. 2013 Nov 12;8(11):e80533. doi: 10.1371/journal.pone.0080533. eCollection 2013. PMID 24265828